CLINICAL TRIAL: NCT00519155
Title: Pilot Study on Safety and Explorative Efficacy of MD05 in Comparison With Open Flap Debridement in Patients Undergoing Periodontal Surgery to Treat Deep Intrabony Defects
Brief Title: Pilot Study on MD05 in Comparison With Open Flap Debridement in Patients Undergoing Periodontal Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Scil Technology GmbH (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Björn Capsius, Scil Technology GmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Scil-MD05-C02; EudraCT-No.: 2006-005883-25
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2008-04

CONDITIONS: Alveolar Bone Loss; Periodontal Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Open flap debridement + MD05
  Interventions: Drug: MD05 and open flap debridement
- 2 (Active Comparator): Open flap debridement
  Interventions: Procedure: Open flap debridement

INTERVENTIONS:
Drug: MD05 and open flap debridement — recombinant human GDF-5 coated onto ß-tricalcium phosphate
  Arms: 1
Procedure: Open flap debridement — Open flap debridement alone
  Arms: 2

SUMMARY:
The purpose of the study is to gain experience of safety and efficacy with MD05 in man in alveolar bone regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring extraction of teeth with advanced intrabony periodontal defects at single rooted teeth without root concavities/furrows located in the maxilla and mandible (maxillary/mandibular premolars, maxillary incisors; presurgery probing depth ≥ 6 mm, intrasurgery defect depth ≥ 4 mm) or located the mesial or distal aspect of mandibular molar teeth without adjacent teeth (excluding defects also involving the furcation area).
* Teeth to be treated must be scheduled for extraction in a treatment plan established by clinicians unrelated to the study.
* Male and female patients, aged 18 - 75 years
* Patients must be non-smokers
* Female patients must be infertile (either sterilized or postmenopausal). If a patient's menopausal status at screening is uncertain, levels of follicle stimulating hormone (FSH) should be determined. Patients with an FSH level > 25 IU/l and absence of menstrual bleeding > 6 months will satisfy the definition of postmenopausal status.
* Patient must provide written informed consent

Exclusion Criteria:

* Women of childbearing potential, pregnant or lactating women
* Participation in another clinical study within 30 days prior to study start
* Previous participation in this study
* Legal incompetence or restricted legal competence
* Alcoholism, drug dependency, smoking
* Acute or chronic infection at the application site
* Known infection with HIV, HBV, or HCV
* Severe allergic rhinitis which requires permanent medication
* Known intolerance of or hypersensitivity to ß-TCP or rhGDF?5
* Presence of local or systemic malignant disease or history of local or systemic malignant disease in the past 5 years.
* Patients requiring chemo- or radiotherapy
* Previous or current radiotherapy of the head
* Chronic liver disorder (AST and/or ALT over 2 times upper limit of normal)
* Impaired renal function (creatinine over 1.5 times upper limit of normal)
* Uncontrolled insulin-dependent diabetes mellitus (HbA1c > 7%)
* Clinically relevant symptoms of thyroid dysfunction
* Severe hypertension (RRdiast > 110 mmHg)
* Clinically relevant cardiovascular disease e.g., decompensated cardiac insufficiency, hemodynamically relevant heart valve defects, or myocardial infarction during the last three months
* Systemic bone disease or illness having influence in bone metabolism (e.g. Osteogenesis imperfecta, Paget's disease, Ehlers-Danlos disease, osteomalacia, renal osteodystrophia, hyperparathyroidism)
* Clinically relevant blood coagulation disorder
* Leukopenia < 3.500 leukocytes/µL
* Previous (within last 2 months before screening visit) or current treatment with systemic corticosteroids of more than 5 mg/day prednisone equivalent
* Previous or current therapy with drugs having any influence on bone metabolism such as calcitonin or parathormone (as teriparatid) within the last 6 months before screening visit, bisphosphonates or fluoride at least for 30 days within the last 12 months before screening visit
* Previous (within last 2 months before screening visit) or current treatment with immunosuppressant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-10 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Evidence of regeneration of alveolar bone. | October 2008

SECONDARY OUTCOMES:
Evidence of uncompromised healing. | October 2008

CONTACTS AND LOCATIONS:
Overall Officials: Anton Sculean, Prof., Principal Investigator — Department of Periodontology; Radboud University Medical Center
Locations (1):
- Department of Periodontology, Semmelweis University Budapest, Budapest, Budapest, Hungary